CLINICAL TRIAL: NCT02710383
Title: Biomarker for Cystic Fibrosis: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarker for Cystic Fibrosis
Acronym: BioCyFi
Status: Terminated | Type: Observational
Why Stopped: Study no longer pursued.
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BCF 06-2018
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Chronic Nasal Congestion; Lung Infection; Breathlessness; Clubbing Toes; Meconium Ileus; Failure to Thrive; Pancreatitis
Keywords: Cystic Fibrosis; Biomarker
MeSH Terms: conditions — Dyspnea; Meconium Ileus; Failure to Thrive; Pancreatitis; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants genetically diagnosed with Cystic fibrosis: Participants diagnosed with Cystic fibrosis aged between 2 months and 50 years

SUMMARY:
International, multicenter, observational, longitudinal study to identify biomarker/s for Cystic fibrosis and to explore the clinical robustness, specificity, and long-term variability of these biomarker/s

DETAILED DESCRIPTION:
Cystic fibrosis (CyFi) is a progressive hereditary disease with the prevalence of 1 in 2500. CyFi is an autosomal recessive disease caused by pathogenic variant/s in the CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) gene encoding Cftr protein.

CyFi causes chronic respiratory damage. Pulmonary findings occur already in infancy, which raises questions whether obstruction might be congenital. Thick, sticky mucus clogs the airways, reduces muco-ciliary clearance and leads to problems with breathing and recurrent bacterial (Pseudomonas aeruginosa) infections, which causes over time the formation of scar tissue (fibrosis) and cysts in the lungs.There is no cure for CyFi; however, symptomatic treatment can help relieve symptoms.

The aim of this study is to identify biomarkers for Cystic fibrosis disease and to explore their clinical robustness, specificity, and long-term variability. An ideal biomarker plays an essential role in the early diagnosis, prediction and therapeutic monitoring of a specific disorder.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent is obtained from the participant or the parent/ legal guardian
* The participant is aged between 2 months and 50 years
* The diagnosis of Cystic fibrosis is genetically confirmed by CENTOGENE

EXCLUSION CRITERIA:

* Informed consent is not obtained from the participant or from the parent/ legal guardian
* The participant is younger than 2 months or older than 50 years
* The diagnosis of Cystic fibrosis is not genetically confirmed by CENTOGENE

Ages: 2 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants genetically diagnosed with Cystic fibrosis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of Cystic fibrosis biomarker/s | 36 months
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and long-term variability of Cystic fibrosis biomarker/s | 36 months
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — Centogene GmbH
Locations (5):
- University Hospital Center Mother Teresa, Tirana, Albania
- Department of Molecular and Medical Genetics, Tbilisi State Medical University, Tbilisi, Georgia
- Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala, India
- Department of Pediatric Gastroenterology and Hepatology, The Children's Hospital and Institute of Child Health, Lahore, Pakistan
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided